CLINICAL TRIAL: NCT01334411
Title: Identifying Good and Poor Surgical Behaviour in the Danish Operating Room
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Lene Spanager, Danish Institute for Medical Simulation, Herlev Hospital
Other Study IDs: NTS-1-LS
Record Dates: First submitted 2011-04-01; First posted 2011-04-13 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Surgical Behaviour in the Operating Room

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Aim: To identify examples of surgeons good and poor intraoperative behaviours related to safe and efficient surgery.

Methods: Ten observations will undertaken in the operating theatres of Rigshospitalet and Herlev Hospital with the researchers taking field notes. This provides the Ph.d student with empirical background knowledge of observed surgical behaviour as well as an understanding of surgical culture. The knowledge will be used to qualify the interviewguide.

8 semi-structured group interviews and 3 individual interviews will be conducted and tape recorded. The interviews will be led by the Ph.d student with an anesthesia nurse present as a co-moderator. The groups will contain 4 - 12 participants.

The interview guide will be developed with a Scottish behavioural marker system as a framework, drawing upon the literature as well as the observations. It will contain questions regarding leadership, communication, teamwork, situation awareness and decision making to facilitate a discussion about surgeons' good and poor behaviours.

Material: Data will be collected in two hospitals in the capital Region of Denmark, Rigshospitalet and Herlev Hospital. Each hospital will provide four focus groups, one containing consultant surgeons in general surgery, one trainee surgeons, one scrub nurses and one containing a mixture of anesthetists and anesthesia nurses. The two latter focus groups is included to get the perspectives of the surgeons' team members since international studies have demonstrated differences of opinion regarding the perceived quality of teamwork amongst operating theatre staff. This study will be the first to build in the opinions of the team members into a behavioural marker system. 3 individual interviews with surgeons will afterwards conducted in one of the hospitals to get a more in-depth discussion.

Data analysis and statistics: The interviews will be fully transcribed and analysed using qualitative method of systematic text condensation. Power calculations are not relevant in this qualitative study. Accepted guidelines state that the number of participants in each group should range between 5 and 15 and the data are from two large university hospitals receiving different patient categories to ensure a certain representative sample of informants.

ELIGIBILITY:
Inclusion Criteria:

* medical professionals at Rigshospitalet and Herlev Hospital

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The interview informants are health care personell in two Danish Hospitals as described in the project description
Sampling Method: Non-Probability Sample
Dates: Start 2010-09; Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris Ostergaard, M.D, Study Chair — Danish Institute for Medical Simulation
Locations (1):
- Danish Institute for Medical Simulation, Herlev, Denmark

REFERENCES:
- [Derived] Spanager L, Lyk-Jensen HT, Dieckmann P, Wettergren A, Rosenberg J, Ostergaard D. Customization of a tool to assess Danish surgeons non-technical skills in the operating room. Dan Med J. 2012 Nov;59(11):A4526. PMID 23171747